Study title: Functionally-tailored Oral Care Intervention for Community-dwelling

**Older Adults With Dementia and Their Caregivers** 

Identifiers: NCT04238520

**Document date: 02-17-2023** 

## Statistical Analysis Plan

First, descriptive statistics were calculated to describe the characteristics of the study participants at baseline, 4-week follow-up, and 3-month follow-up. Wilcoxon rank-sum tests were used to compare continuous/numeric variables between the control and intervention groups at each visit. Fisher's exact tests were used to compare categorical variables. No adjustments have been made for multiple comparisons. After that, Wilcoxon rank-sum tests were used to compare percent and raw score change in the primary outcomes between baseline and 4 weeks and baseline and 3 months in the study and control groups.